CLINICAL TRIAL: NCT03152084
Title: DAPASALT: An Open Label, Phase IV, Mechanistic, Three-Arm Study to Evaluate the Natriuretic Effect of 2-Week Dapagliflozin Treatment in Type 2 Diabetes Mellitus Patients With Either Preserved or Impaired Renal Function and Non-Diabetics With Impaired Renal Function
Brief Title: The Study Will Evaluate Average 24-hr Sodium Excretion During Dapagliflozin Treatment in Patients With Type 2 Diabetes Mellitus With Preserved or Impaired Renal Function or Non-diabetics With Impaired Renal Function.
Acronym: DAPASALT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1690C00049; 2016-002961-79 (EudraCT Number)
Record Dates: First submitted 2017-04-18; First posted 2017-05-12 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 2; Kidney Function Tests
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): T2DM subjects with an eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2 at the Screening Visit.
  Interventions: Drug: Dapagliflozin
- Arm 2 (Experimental): T2DM subjects with an eGFR (CKD-EPI) between >90 and ≤130 mL/min/1.73m2 for patients aged 59 or younger, between >85 and ≤130 mL/min/1.73m2 for patients aged 60 to 69, and between >75 and ≤130 mL/min/1.73m2 for patients aged 70 or older at the Screening Visit.
  Interventions: Drug: Dapagliflozin
- Arm 3 (Experimental): Non-diabetic subjects with an eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2 at the Screening Visit.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — The study consists of a 2-week, open label, dapagliflozin (10mg) treatment period.

SUMMARY:
The purpose of this study is to evaluate how dapagliflozin mechanism of action is impacted by Type 2 Diabetes Mellitus status and kidney function

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Female and/or male aged between 18 years and ≤80 years
* In the diabetic arms - a diagnosis of T2DM with HbA1c ≥6.5% (≥48 mmol/mol) and <10% (<86 mmol/mol); and eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2 or between >90 and ≤130 mL/min/1.73m2 for patients aged 59 years or younger, between >85 and ≤130 mL/min/1.73m2 for patients aged 60 to 69 years, and between >75 and ≤130 mL/min/1.73m2 for patients aged 70 years or older at the Screening Visit (Visit 1)
* In the non-diabetic arm, HbA1c <6.5% (<48 mmol/mol) and an eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2 at the Screening Visit (Visit 1)
* Patient specific optimal antihypertensive dose of an angiotensin receptor blocker at least 6 weeks before study treatment
* In the diabetic arm (Group 2) an appropriate stable dose of metformin, or sulphonylurea, or metformin+sulphonylurea as anti-diabetic therapy for the last 12 weeks before study treatment
* Stable urinary sodium excretion on 2 successive 24-hr urinary sodium excretion measurements.
* In the diabetic arm with impaired renal function (Group 1), a stable insulin dosing (intermediate, long-acting, premixed insulin, basal bolus insulin) for the last 12 weeks prior to Visit 4 (Day 1), as judged by the Investigator. Metformin or sulphonylurea, or metformin+sulphonylurea together with insulin would be accepted, but is not mandatory. If used, stable dose of metformin or sulphonylurea, or metformin+sulphonylurea as anti-diabetic therapy for the last 12 weeks prior to Visit 4 (Day 1) is required.

Exclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus
* Any of the following cardiovascular/vascular diseases within 3 months prior to signing the consent; myocardial infarction, cardiac surgery or revascularization, unstable angina, unstable heart failure, heart failure NYHA Class IV, transient ischemic attack or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia
* Symptoms/complaints suggestive of established neurogenic bladder and/or incomplete bladder emptying
* History of bladder cancer, diagnosis of polycystic kidney disease, history or current lupus nephritis or unstable or rapidly progressing renal disease
* UACR >1000 mg/g at screening
* Current/chronic use of the following medications: any anti-diabetic medication with the exception of metformin, sulphonylurea, angiotensin converting enzyme inhibitors, insulin (insulin only allowed in Group 1), oral glucocorticoids, non-steroidal anti-inflammatory drugs, immune suppressants, chemotherapeutics, antipsychotics, tricyclic antidepressants and monoamine oxidase inhibitors
* Receiving immunosuppressive or other immunotherapy for primary or secondary renal disease within 6 months prior to screening
* Current treatment or treatment within the last 2 weeks prior to screening with diuretics including loop diuretics, thiazides, and mineralocorticoid antagonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (2):
  - Research Site, Almelo
  - Research Site, Amsterdam
- Sweden (2):
  - Research Site, Örebro
  - Research Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Scholtes RA, Muskiet MHA, van Baar MJB, Hesp AC, Greasley PJ, Hammarstedt A, Karlsson C, Hallow KM, Danser AHJ, Heerspink HJL, van Raalte DH. The Adaptive Renal Response for Volume Homeostasis During 2 Weeks of Dapagliflozin Treatment in People With Type 2 Diabetes and Preserved Renal Function on a Sodium-Controlled Diet. Kidney Int Rep. 2022 Mar 4;7(5):1084-1092. doi: 10.1016/j.ekir.2022.02.023. eCollection 2022 May. PMID 35570989
- [Derived] Scholtes RA, Muskiet MHA, van Baar MJB, Hesp AC, Greasley PJ, Karlsson C, Hammarstedt A, Arya N, van Raalte DH, Heerspink HJL. Natriuretic Effect of Two Weeks of Dapagliflozin Treatment in Patients With Type 2 Diabetes and Preserved Kidney Function During Standardized Sodium Intake: Results of the DAPASALT Trial. Diabetes Care. 2021 Feb;44(2):440-447. doi: 10.2337/dc20-2604. Epub 2020 Dec 14. PMID 33318125
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00049&attachmentIdentifier=be370583-b4a1-4b70-beb9-36494cdc972e&fileName=D1690C00049_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00049&attachmentIdentifier=c44b2c01-34f0-4182-ab6f-d195ab6b4d61&fileName=D1690C00049_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 12-Jul-2017 and 20-Mar-2020. Patients who met all the inclusion and none of the exclusion criteria were enrolled in the study.
Pre-assignment Details: All study assessments were performed as per the schedule of assessment. No patients in Group 1 were enrolled into the Run-in set due to failure to meet inclusion exclusion criteria, screen failure, or other reasons. Due to unsatisfactory recruitment rate, it was decided that no more Group 1 patients would be enrolled in the study. Group 1 included type 2 diabetes mellitus (T2DM) patients with impaired kidney function and were to receive oral dose of dapagliflozin 10 mg/day from Day 1 to Day 14.
Groups:
- Group 2: Type 2 diabetes mellitus (T2DM) patients with preserved kidney function received oral dose of dapagliflozin 10 mg/day from Day 1 to Day 14, following which they entered Follow-up Period from Day 15 to Day 19.
- Group 3: Non-diabetic patients with impaired kidney function received oral dose of dapagliflozin 10 mg/day from Day 1 to Day 14, following which they entered Follow-up Period from Day 15 to Day 19.
Period: Overall Study
Arm/Group | Group 2 | Group 3
Started | 17 | 7
Completed | 17 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set: All patients who received at least one dose of study drug and had data from at least one post-dose safety assessment available were included in the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 2 | Group 3 | Total
Number analyzed (Participants) | 17 | 7 | 24
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 80 years | 17 | 7 | 24
  >=80 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Sodium Excretion From Baseline to Start of Treatment
Description: Change in 24-hour sodium excretion during dapagliflozin treatment between baseline and average of Days 2 to 4 within each study group in patients with T2DM with preserved kidney function and in non-diabetics with impaired kidney function was assessed.
Time Frame: From baseline (Day -3 to Day -1) to start of treatment (Day 2 to Day 4)
Population: Evaluable patient set: all patients who dispensed at least one dose of study drug. It excluded primary efficacy variable data which may have been affected by protocol deviations as determined by medical monitor or agreed by study team. For Group 3, early termination of the study resulted in 6 evaluable patients. Due to insufficient number of patients recruited, no statistical conclusions were derived, and no confidence intervals or p-values are presented.
Measure: Median (Full Range); unit: mmol/24 hour
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 15 | 6
mmol/24 hour | -5.33 [-53.667 to 44.000] | -27.67 [-69.334 to 13.334]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.4462, Mixed Models Analysis — Start of treatment vs baseline; Least square mean = -5.21, 95% CI 2-sided [-19.542 to 9.120]

2. Secondary Outcome: Change in 24-hour Sodium Excretion From Baseline to End of Treatment and From End of Treatment to Follow-up
Description: Average change in 24-hour sodium excretion from average baseline values to average end of treatment values (Day 12 to 14); and from average end of treatment values (Day 12 to 14) to average values during follow-up (Day 15 to 17).
Time Frame: From baseline (Day -3 to Day -1) to end of treatment (Day 12 to 14); and from end of treatment (Day 12 to 14) to follow-up (Day 15 to 17)
Population: as for outcome 1
Measure: Median (Full Range); unit: mmol/24 hour
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 15 | 6
mmol/24 hour
  End of treatment vs baseline | 2.67 [-64.000 to 143.167] | -23.83 [-107.000 to 0.667]
  Follow-up vs end of treatment | 1.33 [-135.334 to 25.000] | 6.17 [-70.333 to 20.333]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.7842, Mixed Models Analysis — End of treatment vs baseline; Least square mean = 3.69, 95% CI 2-sided [-24.817 to 32.195]
Statistical Analysis 2: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0581, Regression, Linear — Follow-up vs End of treatment; Least square mean = -16.72, 95% CI 2-sided [-34.109 to 0.664]

3. Secondary Outcome: Change in 24-hour Glucose Excretion From Baseline to Start of Treatment
Description: Average change in 24-hour glucose excretion from average baseline values to average start of treatment values (Day 2 to 4).
Time Frame: From baseline (Day -3 to Day -1) to start of treatment (Day 2 to 4)
Population: Evaluable patient set: all patients who dispensed at least one dose of study drug. Due to insufficient number of patients recruited, no statistical conclusions were derived, and no confidence intervals or p-values are presented for Group 3.
Measure: Median (Full Range); unit: mmol/24 hour
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 15 | 5
mmol/24 hour | 302.61 [191.472 to 635.726] | 43.93 [12.050 to 132.333]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p < 0.0001, Mixed Models Analysis — Start of treatment vs baseline; Least square mean = 344.85, 95% CI 2-sided [272.785 to 416.905]

4. Secondary Outcome: Change in 24-hour Glucose Excretion From Baseline to End of Treatment
Description: Average change in 24-hour glucose excretion from average baseline values to average end of treatment values (Day 12 to 14)
Time Frame: From baseline (Day -3 to Day -1) to end of treatment (Day 12 to 14)
Population: as for outcome 3
Measure: Median (Full Range); unit: mmol/24 hour
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 15 | 4
mmol/24 hour | 283.40 [155.876 to 762.801] | 29.88 [15.450 to 113.300]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p < 0.0001, Mixed Models Analysis — End of treatment vs baseline; Least square mean = 311.30, 95% CI 2-sided [224.528 to 398.064]

5. Secondary Outcome: Change in 24-hour Glucose Excretion From End of Treatment to Follow-up
Description: Average change in 24-hour glucose excretion from average end of treatment values (Day 12 to 14) to average values during follow-up (Day 15 to 17).
Time Frame: From end of treatment (Day 12 to 14) to follow-up (Day 15 to 17)
Population: as for outcome 3
Measure: Median (Full Range); unit: mmol/24 hour
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 15 | 5
mmol/24 hour | -168.43 [-376.561 to -107.596] | -37.02 [-74.733 to -10.584]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p < 0.0001, Regression, Linear — Follow-up vs end of treatment; Least square mean = -203.07, 95% CI 2-sided [-235.983 to -170.162]

6. Secondary Outcome: Change in Mean 24-hour Systolic Blood Pressure From Baseline to Start of Treatment
Description: Change in mean 24-hour systolic blood pressure from baseline to start of treatment (Day 4)
Time Frame: From baseline (Day -1) to start of treatment (Day 4)
Population: as for outcome 3
Measure: Median (Full Range); unit: mmHg
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 13 | 6
mmHg | -5.4810 [-13.6610 to 5.6100] | -8.9730 [-24.6570 to 2.7210]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0047, Mixed Models Analysis — Start of treatment vs baseline; Least square mean = -5.2658, 95% CI 2-sided [-8.5459 to -1.9856]

7. Secondary Outcome: Change in Mean 24-hour Systolic Blood Pressure From Baseline to End of Treatment
Description: Change in mean 24-hour systolic blood pressure from baseline to end of treatment (Day 13).
Time Frame: From baseline (Day -1) to end of treatment (Day 13)
Population: as for outcome 3
Measure: Median (Full Range); unit: mmHg
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 12 | 6
mmHg | -5.9385 [-16.0060 to 0.9160] | -10.3290 [-23.4160 to 16.2160]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0003, Mixed Models Analysis — End of treatment vs baseline; Least square mean = -7.0987, 95% CI 2-sided [-10.0379 to -4.1595]

8. Secondary Outcome: Change in Mean 24-hour Systolic Blood Pressure From End of Treatment to End of Follow-up
Description: Change in mean 24-hour systolic blood pressure from end of treatment (Day 13) to end of follow-up (Day 18).
Time Frame: From end of treatment (Day 13) to end of follow-up (Day 18)
Population: as for outcome 3
Measure: Median (Full Range); unit: mmHg
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 11 | 5
mmHg | 2.5140 [-10.3420 to 8.4590] | -2.6590 [-16.3110 to 7.4680]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.5592, Regression, Linear — Follow-up vs end of treatment; Least square mean = 0.7287, 95% CI 2-sided [-1.9894 to 3.4468]

9. Secondary Outcome: Change in Plasma Volume From Baseline to Start of Treatment
Description: Change in plasma volume from baseline to start of treatment (Day 4).
Time Frame: From baseline (Day 1) to start of treatment (Day 4)
Population: as for outcome 3
Measure: Median (Full Range); unit: Litres
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 13 | 3
Litres | -0.1440 [-1.7819 to 2.6385] | -0.1139 [-2.0340 to 0.0232]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.9288, Mixed Models Analysis — Start of treatment vs baseline; Least square mean = 0.0315, 95% CI 2-sided [-0.7274 to 0.7904]

10. Secondary Outcome: Change in Plasma Volume From Baseline to End of Treatment
Description: Change in plasma volume from baseline to end of treatment (Day 14).
Time Frame: From baseline (Day 1) to end of treatment (Day 14)
Population: as for outcome 3
Measure: Median (Full Range); unit: Litres
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 11 | 1
Litres | -0.2122 [-2.8346 to 1.1073] | 2.0557 [2.0557 to 2.0557]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.1659, Mixed Models Analysis — End of treatment vs baseline; Least square mean = -0.4318, 95% CI 2-sided [-1.0761 to 0.2125]

11. Secondary Outcome: Change in Plasma Volume From End of Treatment to End of Follow-up
Description: Change in plasma volume from end of treatment (Day 14) to end of follow-up (Day 18).
Time Frame: From end of treatment (Day 14) to end of follow-up (Day 18)
Population: as for outcome 3
Measure: Median (Full Range); unit: Litres
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 12 | 0
Litres | 0.6464 [-1.5016 to 1.6410] |
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0190, Regression, Linear — Follow-up vs end of treatment; Least square mean = 0.4755, 95% CI 2-sided [0.0963 to 0.8548]

12. Secondary Outcome: Change in Extracellular Volume From Baseline to Start of Treatment
Description: Change in extracellular volume from baseline to start of treatment (Day 4).
Time Frame: From baseline (Day 1) to start of treatment (Day 4)
Population: as for outcome 3
Measure: Median (Full Range); unit: Litres
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 14 | 6
Litres | -0.5783 [-2.7027 to 0.7959] | -0.4553 [-1.3758 to 0.2282]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0157, Mixed Models Analysis — Start of treatment vs baseline; Least square mean = -0.6713, 95% CI 2-sided [-1.1914 to -0.1511]

13. Secondary Outcome: Change in Extracellular Volume From Baseline to End of Treatment
Description: Change in extracellular volume from baseline to end of treatment (Day 14).
Time Frame: From baseline (Day 1) to end of treatment (Day 14)
Population: as for outcome 3
Measure: Median (Full Range); unit: Litres
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 13 | 6
Litres | 0.1248 [-1.4948 to 0.9852] | -0.1427 [-0.6101 to 1.0055]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.8700, Mixed Models Analysis — End of treatment vs baseline; Least square mean = -0.0324, 95% CI 2-sided [-0.4631 to 0.3984]

14. Secondary Outcome: Change in Extracellular Volume From End of Treatment to End of Follow-up
Description: Change in extracellular volume from end of treatment (Day 14) to end of follow-up (Day 18).
Time Frame: From end of treatment (Day 14) to end of follow-up (Day 18)
Population: as for outcome 3
Measure: Median (Full Range); unit: Litres
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 13 | 6
Litres | 0.1784 [-0.6507 to 0.9780] | 0.1394 [-0.3045 to 0.9014]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.2446, Regression, Linear — Follow-up vs end of treatment; Least square mean = 0.1718, 95% CI 2-sided [-0.1358 to 0.4795]

15. Secondary Outcome: Change in 24-hour Urine Albumin:Creatinine Ratio (UACR)
Description: Average change in mean 24-hour urine albumin:creatinine ratio (UACR) from average baseline to Day 4; and from average baseline values to average end of treatment values (Day 12 to 14).
Time Frame: From baseline (Day -3 to Day -1) to start of treatment (Day 4); and from baseline (Day -3 to Day-1) to end of treatment (Day 12 to 14)
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/mmol
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 15 | 6
mg/mmol
  Start of treatment vs baseline | -0.07 [-30.750 to 6.700] | -5.83 [-35.300 to 0.300]
  End of treatment vs baseline | -0.04 [-17.250 to 0.737] | -7.28 [-35.733 to 0.467]
  Follow-up vs end of treatment | 0.07 [-0.243 to 51.667] | -0.19 [-2.967 to 6.367]
Statistical Analysis 1: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0023, Mixed Models Analysis — Start of treatment vs baseline; Least square mean = -2.10, 95% CI 2-sided [-3.299 to -0.902]
Statistical Analysis 2: Comparison: Group 2; Test type: Other — Within-group change; p < 0.0001, Mixed Models Analysis — End of treatment vs baseline; Least square mean = -1.59, 95% CI 2-sided [-1.929 to -1.256]
Statistical Analysis 3: Comparison: Group 2; Test type: Other — Within-group change; p = 0.0002, Regression, Linear — Follow-up vs end of treatment; Least square mean = 3.88, 95% CI 2-sided [2.215 to 5.553]

16. Secondary Outcome: Pharmacokinetics of Dapagliflozin on Day 4 and Day 14
Description: Dapagliflozin plasma concentration on Day 4 (pre-dose) and Day 14 (pre-dose, 1h, 2h, 4h post-dose)
Time Frame: At pre-dose (Day 4) and at pre-dose, 1h, 2h, 4h post-dose (Day 14)
Population: Pharmacokinetic analysis set: all patients who were dispensed at least one dose of the study drug and for whom at least one of the plasma concentration samples were available and who had no important protocol deviations judged to impact the analysis of the PK data. Here, number analyzed in each row signifies only the patients with available data that were analyzed for that specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 17 | 7
ng/mL
  Day 4, Pre-dose | 4.58 (134.88) | 19.78 (116.54)
  Day 14, Pre-dose: number analyzed (Participants) | 16 | 6
  Day 14, Pre-dose | 4.54 (46.60) | 15.26 (41.97)
  Day 14, 1 h: number analyzed (Participants) | 16 | 6
  Day 14, 1 h | 57.46 (110.66) | 63.83 (150.41)
  Day 14, 2 h: number analyzed (Participants) | 16 | 6
  Day 14, 2 h | 46.47 (49.30) | 60.41 (140.69)
  Day 14, 4 h: number analyzed (Participants) | 17 | 6
  Day 14, 4 h | 29.71 (47.38) | 47.83 (100.41)

17. Secondary Outcome: Number of Patients With AEs and SAEs
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. SAE is an AE that results in any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, or is a significant medical event.
Time Frame: From Day 1 until Day 18 (Follow-up)
Population: as for baseline characteristics
Measure: Number; unit: Patients
Arm/Group | Group 2 | Group 3
Number analyzed (Participants) | 17 | 7
Patients
  Any AE | 6 | 2
  AEs judged as causally related to dapagliflozin | 4 | 0
  AEs leading to death | 0 | 0
  SAEs (including outcomes = death) | 0 | 0
  SAEs causally related to dapagliflozin | 0 | 0
  AEs leading to permanent discontinuation of dapagliflozin | 0 | 0
  SAEs leading to permanent discontinuation of dapagliflozin | 0 | 0
  Hypoglycaemia AEs | 0 | 0
  Hypoglycaemia AEs leading to permanent discontinuation of dapagliflozin | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 until Day 18 (FU)
Description: SAEs and non-SAEs are reported for the Safety Set which comprised of all patients who received at least one dose of study drug and who had data from at least one post-dose safety assessment available.
Arm/Group | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/7
Other Adverse Events (participants affected / at risk) | 6/17 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 2 (N=17) | Group 3 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Genital infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely closed due to unsatisfactory recruitment rate. Of 5 patients enrolled in the Group 1, none were enrolled into the Run-in set due to failure to meet inclusion/exclusion criteria, screen failure, withdrawal or other reason and hence it was decided that no more Group 1 patients would be enrolled in the study. In Group 2 and 3, 17 and 7 patients received the investigational product and completed the study, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results are Sponsor's intellectual property and PIs cannot present or publish results without prior Sponsor approval.

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03152084/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03152084/SAP_001.pdf